CLINICAL TRIAL: NCT04185441
Title: National, Multicenter, Randomized, Double-blind, Double-dummy, Phase III Clinical Trial to Evaluate the Efficacy and Safety of Tanzânia Association in the Treatment of Erectile Dysfunction Associated With Benign Prostatic Hyperplasia
Brief Title: Efficacy and Safety of Tanzânia Association in the Treatment of Erectile Dysfunction Associated With Benign Prostatic Hyperplasia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: EMS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EMS0119 - TANZÂNIA
Record Dates: First submitted 2019-12-02; First posted 2019-12-04 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Erectile Dysfunction; Benign Prostatic Hyperplasia
Keywords: Erectile Dysfunction; Benign Prostatic Hyperplasia
MeSH Terms: conditions — Erectile Dysfunction; Prostatic Hyperplasia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TANZÂNIA (Experimental): The study is double-dummy. The patient must take 2 pills, as follow:
  1 capsule Tanzânia association, oral, once a day, and
  1 tablet tamsulosin placebo, oral, once a day.
  Interventions: Drug: Tanzânia association; Other: Omnic Ocas placebo
- Omnic Ocas (Active Comparator): The study is double-dummy. The patient must take 2 pills, as follow:
  1 tablet Omnic Ocas, oral, once a day, and
  1 capsule Tanzânia association placebo, oral, once a day.
  Interventions: Drug: Omnic Ocas; Other: Tanzânia association placebo

INTERVENTIONS:
Drug: Tanzânia association — Tanzânia association capsule
  Arms: TANZÂNIA
Drug: Omnic Ocas — Tamsulosin 0,4 mg
  Arms: Omnic Ocas
Other: Omnic Ocas placebo — Tamsulosin placebo
  Arms: TANZÂNIA
Other: Tanzânia association placebo — EMS association placebo
  Arms: Omnic Ocas

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Tanzânia association in adults with erectile dysfunction associated with Benign Prostatic Hyperplasia.

ELIGIBILITY:
Inclusion Criteria:

* Ability to confirm voluntary participation and agree to all trial purposes by signing and dating the informed consent forms;
* Male participants aged 18 years or more;
* Sexually active participants with a defined partner who have averaged 1 attempt at sexual intercourse per week in the past month;
* Diagnosis of Benign Prostatic Hyperplasia;
* Diagnosis of erectile dysfunction;
* Patients with score between 6 and 25 points in the erectile function questionnaire;
* IPSS (International Prostate Symptom Score) greater or equal to 8 points;

Exclusion Criteria:

* Known hypersensitivity to the formula components used during the clinical trial;
* History of alcohol and/or substance abuse within 2 years;
* Diagnosis of other diseases or conditions in the urinary tract, including but not limited to: cancer, neurogenic bladder; urinary incontinence, recurrent infection, urethral stricture, bacterial prostatitis;
* Clinical evidence of prostate cancer;
* Hypogonadism or absent sexual desire;
* Severe psychiatric or psychosocial disorders;
* Primary erectile dysfunction;
* Polyneuropathy, neurodegenerative diseases, trauma or spinal cord injuries, central nervous system tumors or other conditions that may affect erections;
* Anatomical penile deformation that can significantly impair erection, including but not limited to: angulation, cavernous fibrosis, Peyronie's disease.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 295 (Actual)
Dates: Start 2021-03-14 (Actual); Primary Completion 2023-10-10 (Actual); Study Completion 2024-07-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in erectile function questionnaire. | 8 weeks
  The erectile function questionnaire score ranges from 1 to 30 points. The lower the score, the higher the degree of erectile dysfunction.

SECONDARY OUTCOMES:
Incidence and severity of adverse events recorded during the study. | 10 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Allergisa, Campinas, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No